CLINICAL TRIAL: NCT00988143
Title: Immunogenicity and Safety Among Children and Adults of the 2009-2010 Trivalent Influenza Vaccine, 2008-2009 Trivalent Influenza Vaccine, and Quadrivalent Influenza Vaccine (Intramuscular Route)
Brief Title: A Study of Influenza Virus Vaccines in Children and Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC43; UTN: U1111-1111-5427 (Other: WHO)
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Results first posted 2013-12-12 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-11

CONDITIONS: Influenza
Keywords: Influenza; Trivalent Influenza Virus Vaccine; Quadrivalent Influenza Virus Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Study Group 1 (Experimental): Participants will receive the 2009-2010 Trivalent Influenza Vaccine (TIV) (Pediatric dose have no preservatives)
  Interventions: Biological: 2009-2010 Trivalent Influenza Virus Vaccine
- Study Group 2 (Active Comparator): Participants will receive the 2008-2009 Trivalent Influenza Vaccine (TIV)
  Interventions: Biological: 2008-2009 Trivalent Influenza Virus Vaccine
- Study Group 3 (Active Comparator): Participants will receive the Quadrivalent Influenza Vaccine (QIV)
  Interventions: Biological: Quadrivalent Influenza Virus Vaccine

INTERVENTIONS:
Biological: 2009-2010 Trivalent Influenza Virus Vaccine — 0.25 mL, Intramuscular (participants at 6 to 35 months of age - Pediatric Dose); Others 0.5 mL, Intramuscular.
  Other Names: Fluzone®
  Arms: Study Group 1
Biological: 2008-2009 Trivalent Influenza Virus Vaccine — 0.25 mL, Intramuscular; 0.5 mL, Intramuscular.
  Other Names: Fluzone®
  Arms: Study Group 2
Biological: Quadrivalent Influenza Virus Vaccine — 0.5 mL, Intramuscular
  Arms: Study Group 3

SUMMARY:
The purpose of this study is to describe the immunogenicity of the prototype Quadrivalent Influenza Vaccine (QIV) compared with the 2009-2010 Trivalent Influenza Vaccine (TIV) and the 2008-2009 TIV among children and adults.

Primary Objective:

To describe the immunogenicity of the prototype Quadrivalent Influenza Vaccine (QIV) compared with the 2009-2010 Trivalent Influenza Vaccine (TIV) and the 2008-2009 TIV among adults.

Observational Objectives:

* To describe the safety of the 2009-2010 TIV among subjects ≥6 months to <5 years, 18-60 years, and ≥ 61 years of age, and to describe the safety of 2008-2009 TIV and prototype QIV Fluzone® vaccines among subjects 18-60 years and ≥ 61 years of age.
* To describe the immunogenicity of the 2009-2010 TIV vaccine among subjects ≥6 months to <5 years, 18-60 years, and ≥61 years of age, and to describe the immunogenicity of 2008-2009 TIV and prototype QIV vaccines among subjects 18-60 years and ≥61 years of age.

ELIGIBILITY:
Inclusion Criteria :

* Subject is ≥ 6 months to < 5 years of age or 18 years of age or older on the day of inclusion.
* Parent/legal guardian (if the subject is ≥ 6 months to < 5 years of age) or adult subject (if 18 years of age or older) is willing and able to attend scheduled visits and to comply with the study procedures during the entire duration of the study.
* Subject in reasonably good health as assessed by the Investigator.
* Parent/legal guardian (if the subject is ≥ 6 months to < 5 years of age) or adult subject (if 18 years of age or older) is willing and able to give informed consent.
* For subjects ≥ 6 months to < 5 years of age: subject was born at full term of pregnancy (≥ 37 weeks) with a birth weight ≥ 2.5 kg (5.5 lbs).
* For a woman, inability to bear a child or negative serum/urine pregnancy test, if applicable.

Exclusion Criteria :

For all subjects:

* History of allergy to egg proteins, chicken proteins, or one of the constituents of the vaccine, such as thimerosal or formaldehyde.
* History of serious adverse reaction to any influenza vaccine.
* Laboratory-confirmed influenza infection or vaccination against influenza in the six months preceding enrollment in the study.
* Any vaccination scheduled between Visit 1 and Visit 2 or Visit 3.
* Participation in any other interventional drug or vaccine trial during participation in this study.
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination.
* Any condition that in the opinion of the Investigator would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine.
* Prior personal history of Guillain-Barré syndrome.

For subjects > 6 months to < 5 years of age:

* Known or suspected impairment of immunologic function or receipt of immunosuppressive therapy or immunoglobulin since birth.
* Personal or immediate family history of congenital immune deficiency.
* Developmental delay, neurologic disorder, or seizure disorder.
* Chronic medical, congenital, or developmental disorder.
* Known HIV-positive mother.

For subjects 18 years of age and older:

* Immunocompromising condition; immunosuppressive therapy (including systemic steroid use for two weeks or more); cancer chemotherapy or radiation therapy at the time of enrollment, planned during the period of this study, or at any time within the past six months.
* Diabetes mellitus requiring pharmacological control.
* Person deprived of freedom by an administrative or court order (having legal or medical guardian).
* For women of childbearing potential, a positive urine pregnancy test, breast feeding, or not using a medically approved and reliable form of contraception (oral contraceptives or double barrier method) for the duration of the trial.
* Current use of alcohol or recreational drugs that may interfere with the subject's ability to comply with trial procedures.
* Any subject with the following conditions is not eligible for enrollment. However, the subject may be enrolled subsequently if the condition has resolved and enrollment is still ongoing and the subject meets all other inclusion/exclusion criteria:

  * An acute illness with or without fever in the 72 hours preceding enrollment in the trial.
  * Clinically significant findings in vital signs or review of systems (Investigator judgment).
  * Received any vaccinations within the preceding 14 days.
  * Participation in any other interventional clinical trial within 30 days prior to enrollment.
  * Receipt of blood or blood products within the three months preceding enrollment in the study.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (4):
- United States (4):
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Jefferson Hills, Pennsylvania
  - Norfolk, Virginia

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 01 October through 05 November 2009 in 4 clinical centers in the US.
Pre-assignment Details: A total of 600 participants who met all the inclusion criteria and none of the exclusion criteria were enrolled, randomized and vaccinated in the study.
Groups:
- Study Group 1 (2009-2010 TIV): Participants received the 2009-2010 Trivalent Influenza Vaccine (Pediatric dose with no preservatives)
- Study Group 2 (2008-2009 TIV): Participants received the 2008-2009 Trivalent Influenza Vaccine
- Study Group 3 (QIV): Participants received the Quadrivalent Influenza Vaccine
Period: Overall Study
Arm/Group | Study Group 1 (2009-2010 TIV) | Study Group 2 (2008-2009 TIV) | Study Group 3 (QIV)
Started | 220 | 190 | 190
Completed | 220 | 190 | 190
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Group 1 (2009-2010 Trivalent Influenza Vaccine): Participants received the 2009-2010 Trivalent Influenza Vaccine (TIV)
- Study Group 2 (2008-2009 Trivalent Influenza Vaccine): Participants received the 2008-2009 Trivalent Influenza Vaccine (TIV)
- Study Group 3 (Quadrivalent Influenza Vaccine): Participants received the Quadrivalent Influenza Vaccine (QIV)
- Total: Total of all reporting groups
Arm/Group | Study Group 1 (2009-2010 Trivalent Influenza Vaccine) | Study Group 2 (2008-2009 Trivalent Influenza Vaccine) | Study Group 3 (Quadrivalent Influenza Vaccine) | Total
Number analyzed (Participants) | 220 | 190 | 190 | 600
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 0 | 0 | 30
  Between 18 and 65 years | 127 | 135 | 123 | 385
  >=65 years | 63 | 55 | 67 | 185
Age Continuous [Mean (Standard Deviation); unit: Years] | 47.8 (24.9) | 54.9 (17.5) | 56.7 (17.2) | 52.9 (20.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 124 | 130 | 398
  Male | 76 | 66 | 60 | 202
Region of Enrollment [Number; unit: Participants]
  United States | 220 | 190 | 190 | 600

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactions Following Vaccination With Quadrivalent Influenza Vaccine or Fluzone® Trivalent Influenza Vaccines.
Description: Solicited injection site reactions (6-23 Months): Tenderness, Redness and Swelling; Solicited systemic reactions: Fever, Abnormal crying, Drowsiness, Loss of appetite, Vomiting and Irritability Grade 3 Tenderness: cries when injected limb is moved; Redness and Swelling: ≥5 cm; Fever: >103.1°F; Abnormal crying: >3 hours; Drowsiness: Sleeping most of the time; Loss of appetite: refuses ≥3 feeds/meals; Vomiting: ≥6 episodes/24 hours; Irritability: inconsolable.
  (24-59 Months): Pain, Redness and Swelling; Fever, Headache, Malaise and Myalgia. Grade 3: Pain, Incapacitating; Redness and Swelling: ≥5 cm; Fever: >102.1°F, Headache, Malaise and Myalgia: Significant, prevents daily activity.
  (Adults): Pain, Redness, Induration, and Ecchymosis; Fever, Headache, Malaise, Myalgia and Shivering.
  Grade 3: Pain: significant, prevents daily activities; Redness, Swelling, Induration and Ecchymosis: >10 cm; Fever >102.1°F; Headache, Malaise, Myalgia & Shivering: Significant, prevents daily activity.
Time Frame: Day 0 up to 7 days post-vaccination
Population: Solicited injection site and systemic reactions were assessed in all randomized and vaccinated participants, safety population.
Measure: Number; unit: Participants
Arm/Group | Study Group 1 (2009-2010 Trivalent Influenza Vaccine) | Study Group 2 (2008-2009 Trivalent Influenza Vaccine) | Study Group 3 (Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 220 | 190 | 190
Participants
  Injection site Tenderness (15, 0, 0) | 4 | 0 [0 to 0] | 0 [0 to 0]
  Grade 3 Injection site Tenderness (15, 0, 0) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Injection site Pain (205, 190, 190) | 105 | 82 [0 to 0] | 90 [0 to 0]
  Grade 3 Injection site Pain (206, 190, 190) | 1 | 0 [0 to 0] | 1 [0 to 0]
  Injection site Erythema (220, 190, 190) | 7 | 3 [0 to 0] | 2 [0 to 0]
  Grade 3 Injection site Erythema (220, 190, 190) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Injection site Swelling (220, 190, 190) | 10 | 2 [0 to 0] | 1 [0 to 0]
  Grade 3 Injection site Swelling (220, 190, 190) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Injection site Induration (190, 190, 190) | 3 | 1 [0 to 0] | 1 [0 to 0]
  Grade 3 Injection site Induration (190, 190, 190) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Injection site Ecchymosis (190, 190, 190) | 1 | 1 [0 to 0] | 1 [0 to 0]
  Grade 3 Injection site Ecchymosis (190, 190, 190) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Fever (220, 190, 190) | 2 | 1 [0 to 0] | 0 [0 to 0]
  Grade 3 Fever (220, 190, 190) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Vomiting (15, 0, 0) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Grade 3 Vomiting (15, 0, 0) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Malaise (205, 190, 190) | 30 | 23 [0 to 0] | 20 [0 to 0]
  Grade 3 Malaise (205, 190, 190) | 3 | 1 [0 to 0] | 2 [0 to 0]
  Appetite lost (15, 0, 0) | 1 | 0 [0 to 0] | 0 [0 to 0]
  Grade 3 Appetite lost (15, 0, 0) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Drowsiness (15, 0, 0) | 4 | 0 [0 to 0] | 0 [0 to 0]
  Grade 3 Drowsiness (15, 0, 0) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Crying abnormal (15, 0, 0) | 1 | 0 [0 to 0] | 0 [0 to 0]
  Grade 3 Crying abnormal (15, 0, 0) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Headache (205, 189, 190) | 35 | 34 [0 to 0] | 30 [0 to 0]
  Grade 3 Headache (205, 189, 190) | 1 | 0 [0 to 0] | 1 [0 to 0]
  Irritability (15, 0, 0) | 5 | 0 [0 to 0] | 0 [0 to 0]
  Grade 3 Irritability (15, 0, 0) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Myalgia (205, 190, 190) | 50 | 32 [0 to 0] | 45 [0 to 0]
  Grade 3 Myalgia (205, 190, 190) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Shivering (190, 190, 190) | 10 | 6 [0 to 0] | 5 [0 to 0]
  Grade 3 Shivering (190, 190, 190) | 0 | 0 [0 to 0] | 0 [0 to 0]

2. Primary Outcome: Geometric Mean Titers (GMTs) Against Influenza B Strains After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccine in Adult Participants.
Description: Immunogenicity outcomes were assessed in serum samples by Hemagglutination inhibition (HAI) assay. The lower limit of quantitation (LLOQ) was set at the lowest dilution used in the assay, 1/10. Titers below this level were reported as <10.
Time Frame: 21 Days post last vaccination
Population: Geometric mean titers to vaccine B strains were determined in randomized and vaccinated participants, per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Study Group 1 (2009-2010 Trivalent Influenza Vaccine) | Study Group 2 (2008-2009 Trivalent Influenza Vaccine) | Study Group 3 (Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 187 | 188 | 190
Titers
  B/Brisbane/60/2008 (187, 0, 190) | 114 [97.8 to 134] | NA [NA to NA] — B/Brisbane influenza virus antigen not in the vaccine administered to this group | 101 [85.6 to 120]
  B/Florida/04/2006 (0, 188, 190) | NA [NA to NA] — B/Florida influenza virus antigen not in the vaccine administered to this group | 135 [117 to 156] | 155 [133 to 180]

3. Other Pre Specified Outcome: Number of Adult Participants With Seroprotection Against Influenza Vaccine Antigens Following Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccine
Description: Immunogenicity outcomes were assessed in serum samples by HAI assay. The lower limit of quantitation (LLOQ) was set at the lowest dilution used in the assay, 1/10. Titers below this level were reported as <10.
  Seroprotection to vaccine antigens was defined as a pre-vaccination and post-vaccination titer value of titer ≥ 40 (1/dil)
Time Frame: Day 0 (pre-vaccination) and Day 21 post final vaccination
Population: Seroprotection against the influenza vaccine antigens were determined in randomized and vaccinated participants, per-protocol population.
Measure: Number; unit: Participants
Arm/Group | Study Group 1 (2009-2010 Trivalent Influenza Vaccine) | Study Group 2 (2008-2009 Trivalent Influenza Vaccine) | Study Group 3 (Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 187 | 188 | 190
Participants
  A/H1N1, Pre-vaccination (186, 188, 190) | 84 | 77 [23.1 to 33.6] | 81 [0 to 0]
  A/H1N1, Post-vaccination (187, 188, 190) | 168 | 173 [123 to 172] | 176 [0 to 0]
  A/H3N2, Pre-vaccination (186, 187, 190) | 83 | 91 [27.7 to 43.3] | 93 [0 to 0]
  A/H3N2, Post-vaccination (187, 188, 190) | 180 | 177 [271 to 401] | 180 [0 to 0]
  B/Brisbane/60/2008, Pre-vaccination (186, 0, 190) | 80 | NA [0 to 0] — B/Brisbane/60/2008 influenza virus antigen was not in the vaccine administered to this group. | 69 [0 to 0]
  B/Brisbane/60/2008, Post-vaccination (187, 0, 190) | 168 | NA [0 to 0] — B/Brisbane/60/2008 influenza virus antigen was not in the vaccine administered to this group. | 162 [0 to 0]
  B/Florida/04/2006, Pre-vaccination (0, 187, 190) | NA — B/Florida/04/2006 influenza virus antigen was not in the vaccine administered to this group. | 97 [22.8 to 31.1] | 89 [0 to 0]
  B/Florida/04/2006, Post-vaccination (0, 187, 190) | NA — B/Florida/04/2006 influenza virus antigen was not in the vaccine administered to this group. | 174 [84.0 to 111] | 175 [0 to 0]

4. Other Pre Specified Outcome: Geometric Mean Titers Against the Influenza Vaccine Antigens After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines in Adult Participants
Description: Immunogenicity outcomes were assessed in serum samples by HAI assay. The lower limit of quantitation (LLOQ) was set at the lowest dilution used in the assay, 1/10. Titers below this level were reported as <10.
Time Frame: 21 Days post last vaccination
Population: Geometric mean titers to influenza vaccine antigens were determined in randomized and vaccinated participants, per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Study Group 1 (2009-2010 Trivalent Influenza Vaccine) | Study Group 2 (2008-2009 Trivalent Influenza Vaccine) | Study Group 3 (Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 187 | 188 | 190
Titers
  A/H1N1, Pre-vaccination (186, 188, 190) | 27.5 [22.8 to 33.0] | 28.4 [23.6 to 34.3] | 27.6 [22.7 to 33.6]
  A/H1N1, Post-vaccination (187, 188, 190) | 145 [122 to 173] | 157 [132 to 187] | 161 [137 to 189]
  A/H3N2, Pre-vaccination (186, 188, 190) | 29.9 [24.0 to 37.2] | 32.7 [25.8 to 41.6] | 38.5 [29.7 to 49.9]
  A/H3N2, Post-vaccination (187, 188, 190) | 302 [250 to 365] | 380 [305 to 472] | 304 [249 to 370]
  B/Brisbane/60/2008, Pre-vaccination (186, 0, 190) | 22.0 [18.5 to 26.2] | NA [NA to NA] — B/Brisbane/60/2008 influenza virus antigen not in the vaccine administered to this group. | 19.9 [16.7 to 23.7]
  B/Brisbane/60/2008, Post-vaccination (187, 0, 190) | 114 [97.8 to 134] | NA [NA to NA] — B/Brisbane/60/2008 influenza virus antigen not in the vaccine administered to this group. | 101 [85.6 to 120]
  B/Florida/04/2006, Pre-vaccination (0, 187, 190) | NA [NA to NA] — B/Florida/04/2006 influenza virus antigen not in the vaccine administered to this group. | 32.6 [27.4 to 38.7] | 27.1 [22.5 to 32.6]
  B/Florida/04/2006, Post-vaccination (0, 187, 190) | NA [NA to NA] — B/Florida/04/2006 influenza virus antigen not in the vaccine administered to this group. | 135 [117 to 156] | 155 [133 to 180]

5. Other Pre Specified Outcome: Number of Adult Participants With Seroconversion to Vaccine Antigens Following Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines
Description: Seroconversion to vaccine antigens was defined as a pre-vaccination titer < 10 (1/dil) and a post-vaccination titer ≥ 40 (1/dil), or a pre-vaccination titer ≥ 10 (1/dil) and a ≥ 4-fold increase in post-vaccination titer.
Time Frame: Day 21 post-vaccination
Population: Seroconversion with respect to vaccine antigens were determined in randomized and vaccinated participants, per-protocol population.
Measure: Number; unit: Participants
Arm/Group | Study Group 1 (2009-2010 Trivalent Influenza Vaccine) | Study Group 2 (2008-2009 Trivalent Influenza Vaccine) | Study Group 3 (Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 187 | 188 | 190
Participants
  A/H1N1 (187, 188, 190) | 103 | 97 [0 to 0] | 112 [0 to 0]
  A/H3N2 (187, 188, 190) | 130 | 120 [0 to 0] | 119 [0 to 0]
  B/Brisbane/60/2008 (187, 0, 190) | 104 | NA [0 to 0] — B/Brisbane/60/2008 influenza virus antigen was not in the vaccine administered to this group. | 101 [0 to 0]
  B/Florida/04/2006 (0, 188, 190) | NA — B/Florida/04/2006 influenza virus antigen was not in the vaccine administered to this group. | 83 [0 to 0] | 110 [0 to 0]

6. Other Pre Specified Outcome: Geometric Mean Titers Against the Influenza Vaccine Antigens After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines in All Study Participants
Description: as for outcome 4
Time Frame: 21 Days post last vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Study Group 1 (2009-2010 Trivalent Influenza Vaccine) | Study Group 2 (2008-2009 Trivalent Influenza Vaccine) | Study Group 3 (Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 215 | 188 | 189
Titers
  A/H1N1, Pre-vaccination (214, 186, 189) | 27.0 [22.8 to 32.1] | 27.8 [23.1 to 33.6] | 25.4 [21.0 to 30.8]
  A/H1N1, Post-vaccination (214, 187, 189) | 153 [131 to 179] | 145 [123 to 172] | 143 [122 to 168]
  A/H3N2, Pre-vaccination (214, 187, 189) | 30.5 [25.1 to 37.2] | 34.6 [27.7 to 43.3] | 37.8 [29.8 to 47.9]
  A/H3N2, Post-vaccination (214, 188, 189) | 285 [244 to 334] | 330 [271 to 401] | 263 [219 to 316]
  B/Brisbane/60/2008, Pre-vaccination (214, 0, 189) | 15.5 [13.4 to 18.0] | NA [NA to NA] — B/Brisbane/60/2008 influenza virus antigen was not in vaccine administered to this group. | 16.2 [13.9 to 18.8]
  B/Brisbane/60/2008, Post-vaccination (215, 0, 189) | 76.7 [66.6 to 88.4] | NA [NA to NA] — B/Brisbane/60/2008 influenza virus antigen was not in vaccine administered to this group. | 75.6 [64.8 to 88.2]
  B/Florida/04/2006, Pre-vaccination (0, 186, 189) | NA [NA to NA] — B/Florida/04/2006 influenza virus antigen was not in vaccine administered to this group. | 26.6 [22.8 to 31.1] | 21.7 [18.3 to 25.7]
  B/Florida/04/2006, Post-vaccination (0, 187, 189) | NA [NA to NA] — B/Florida/04/2006 influenza virus antigen was not in vaccine administered to this group. | 96.5 [84.0 to 111] | 109 [94.5 to 125]

7. Other Pre Specified Outcome: Number of Participants With Seroconversion to Influenza Vaccine Antigens Following Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines
Description: Seroconversion to vaccine antigens were defined as a pre-vaccination titer < 10 (1/dil) and a post-vaccination titer ≥ 40 (1/dil), or a pre-vaccination titer ≥ 10 (1/dil) and a ≥ 4-fold increase in post-vaccination titer.
Time Frame: Day 0 up to 21 days post-vaccination
Population: Seroconversion with respects to influenza vaccine antigens were determined in randomized and vaccinated participants, per-protocol population
Measure: Number; unit: Participants
Arm/Group | Study Group 1 (2009-2010 Trivalent Influenza Vaccine) | Study Group 2 (2008-2009 Trivalent Influenza Vaccine) | Study Group 3 (Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 215 | 188 | 189
Participants
  A/H1N1 Pre-vaccination (214, 186, 189) | 88 | 71 | 70
  A/H1N1 Post-vaccination (213, 186, 189) | 118 | 90 | 112
  A/H3N2 Pre-vaccination (214, 187, 189) | 100 | 94 | 92
  A/H3N2 Post-vaccination (213, 187, 189) | 148 | 119 | 116
  B/Brisbane/60/2008 Pre-vaccination (214, 0, 189) | 57 | NA — B/Brisbane/60/2008 influenza virus antigen was not in the vaccine administered to this group. | 50
  B/Brisbane/60/2008 Post-vaccination (214, 0, 189) | 111 | NA — B/Brisbane/60/2008 influenza virus antigen was not in the vaccine administered to this group. | 99
  B/Florida/04/2006 Pre-vaccination (0, 186, 189) | NA — B/Florida/04/2006 influenza virus antigen was not in the vaccine administered to this group. | 80 | 67
  B/Florida/04/2006 Post-vaccination (0, 186, 189) | NA — B/Florida/04/2006 influenza virus antigen was not in the vaccine administered to this group | 79 | 100

8. Other Pre Specified Outcome: Number of Participants With Seroprotection to Influenza Vaccine Antigens Following Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines
Description: as for outcome 3
Time Frame: Day 0 (pre-vaccination) and Day 21 post final vaccination
Population: Seroprotection to influenza vaccine antigens were determined in randomized and vaccinated participants, per-protocol population
Measure: Number; unit: Participants
Arm/Group | Study Group 1 (2009-2010 Trivalent Influenza Vaccine) | Study Group 2 (2008-2009 Trivalent Influenza Vaccine) | Study Group 3 (Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 215 | 188 | 189
Participants
  A/H1N1, Pre-vaccination (214, 186, 189) | 88 | 71 | 70
  A/H1N1, Post-vaccination (214, 187, 189) | 193 | 168 | 169
  A/H3N2, Pre-vaccination (214, 187, 189) | 100 | 94 | 92
  A/H3N2, Post-vaccination (214, 188, 189) | 209 | 179 | 179
  B/Brisbane/60/2008, Pre-vaccination (214, 0, 189) | 57 | NA — B/Brisbane/60/2008 influenza virus antigen was not in the vaccine administered to this group. | 50
  B/Brisbane/60/2008, Post-vaccination (215, 0, 189) | 172 | NA — B/Brisbane/60/2008 influenza virus antigen was not in the vaccine administered to this group. | 153
  B/Florida/04/2006, Pre-vaccination (0, 186, 189) | NA — B/Florida/04/2006 influenza virus antigen was not in the vaccine administered to this group. | 80 | 67
  B/Florida/04/2006, Post-vaccination (0, 187, 189) | NA — B/Florida/04/2006 influenza virus antigen was not in the vaccine administered to this group. | 164 | 169

9. Primary Outcome: Geometric Mean Titers (GMTs) Against Influenza A Strains After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccine in Adult Participants.
Description: as for outcome 2
Time Frame: 21 Days post last vaccination
Population: Geometric mean titers to vaccine A strains were determined in the per-protocol population. For this outcome, the data for the A/Brisbane/59/2007(A1N1) and A/Uruguay/716/2007(H3N2) antibodies were pooled for participants vaccinated with either 2009-2010 TIV or 2008-2009 TIV and presented in the column for Study Group 1 (2009-2010 TIV).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Study Group 1 (2009-2010 Trivalent Influenza Vaccine) | Study Group 2 (2008-2009 Trivalent Influenza Vaccine) | Study Group 3 (Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 375 | 0 | 190
Titers
  A/Brisbane/59/2007(A1N1) [N = 375, 0, 190] | 151 [134 to 171] |  | 161 [137 to 189]
  A/Uruguay/716/2007(H3N2) [N = 375, 0, 190] | 339 [239 to 392] |  | 304 [249 to 370]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination (Day 0) up to 28 days post-vaccination
Arm/Group | Study Group 1 (2009-2010 Trivalent Influenza Vaccine) | Study Group 2 (2008-2009 Trivalent Influenza Vaccine) | Study Group 3 (Quadrivalent Influenza Vaccine)
Serious Adverse Events (participants affected / at risk) | 0/220 | 0/190 | 2/190
Other Adverse Events (participants affected / at risk) | 105/220 | 84/190 | 91/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Study Group 1 (2009-2010 Trivalent Influenza Vaccine) (N=220) | Study Group 2 (2008-2009 Trivalent Influenza Vaccine) (N=190) | Study Group 3 (Quadrivalent Influenza Vaccine) (N=190)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0/0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0/0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Study Group 1 (2009-2010 Trivalent Influenza Vaccine) (N=220) | Study Group 2 (2008-2009 Trivalent Influenza Vaccine) (N=190) | Study Group 3 (Quadrivalent Influenza Vaccine) (N=190)
Pyrexia (Gastrointestinal disorders) | 2/30 (2) | 0/0 (0) | 0/0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3/30 (3) | 0/0 (0) | 0/0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6/30 (6) | 0/0 (0) | 0/0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2/30 (2) | 0/0 (0) | 0/0 (0)
Headache (Nervous system disorders) | 10/190 (12) | 10 (10) | 5 (5)
Injection site Pain (General disorders) | 105/215 (105) | 82 (82) | 90 (90)
Appetite lost (Metabolism and nutrition disorders) | 1/15 (1) | 0/0 (0) | 0/0 (0)
Drowsiness (Nervous system disorders) | 4/15 (4) | 0/0 (0) | 0/0 (0)
Crying abnormal (Psychiatric disorders) | 1/15 (1) | 0/0 (0) | 0/0 (0)
Irritability (Psychiatric disorders) | 1/15 (1) | 0/0 (0) | 0/0 (0)
Headache (Nervous system disorders) | 35 (35) | 34 (34) | 30 (30)
Malaise (General disorders) | 30 (30) | 23 (23) | 20 (20)
Myalgia (Musculoskeletal and connective tissue disorders) | 50 (50) | 32 (32) | 45 (45)
Shivering (General disorders) | 10/190 (10) | 6 (6) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications